CLINICAL TRIAL: NCT00502372
Title: Nutritional Effect of an Oral Supplement Enriched in Arginine, Glutamine and Leucine Metabolite B-Hydroxy B-Methylbutyrate
Brief Title: Effect of an Oral Supplement Enriched in Amino Acids and the Leucine Metabolite B-hydroxy B-methylbutyrate (HMB)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: VA never granted approval following suspension of enrollment.
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJ93
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer | interventions — Dietary Supplements; Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enriched product, dietary supplement (Experimental): Subjects receiving enriched product compared to an unenriched product
  Interventions: Dietary Supplement: Nutritional Supplement/Amino acids and HMB; Dietary Supplement: Juven
- 1 (Active Comparator): Subjects not receiving enriched product
  Interventions: Dietary Supplement: Nutritional Supplement/Amino acids and HMB; Dietary Supplement: Juven

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement/Amino acids and HMB — Subjects will be randomized to receive enriched dietary supplement (Juven) v arginine only (Argenaid) dietary supplement
  Other Names: Juven; Argenaid
Dietary Supplement: Juven — comparison of Juven with arginine only product in wound healing
  Other Names: Argenaid

SUMMARY:
The focus of this study is to look at the role of nutrition in the healing of pressure ulcers. The purpose of this study is to test whether the rate of healing of pressure ulcers is increased in those patients receiving a nutritional supplement of amino acids and the leucine metabolite, B-hydroxy-B-methylbutyrate is enhanced when compared to control patients receiving a supplement containing only one of the proteins in the experimental supplement

DETAILED DESCRIPTION:
Patients who have pressure ulcers Stage II or greater will be randomized to receiving one of two nutritional supplements. One supplement contains arginine and the other contains both arginine,glutamine and leucine metabolites. Pressure ulcers will be measured at study entry and measured biweekly using a standardized tool (PUSH) until the trial is completed or the pressure ulcer has healed.

Inclusion criteria include:

* Stage II or greater pressure ulcer
* Patient consent
* Patients who can drink supplement or receive it by tube
* Patients who are 21 years old or greater

Exclusion criteria include:

* Patients with infected wounds
* Patients with cellulitis, sepsis or osteomyelitis
* Patients with end-organ failure
* Patients with poorly controlled diabetes mellitus (HbA1C>10)
* Patients who cannot tolerate oral or tube feeding

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage II pressure ulcer or greater
2. Patients who consent to participate
3. Patients who can ingest the supplement either orally or per feeding tube
4. Patients who are 21 years of age or older

Exclusion Criteria:

1. Patients with infected wounds
2. Patients with cellulitis, sepsis or osteomyelitis
3. Patients with end-organ failure
4. Patients with poorly controlled diabetes mellitus (HbA1C>10)
5. Patients who cannot tolerate oral or bolus tube feedings

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
PUSH tool score | 8 weeks or healing completed
  The PUSH tool measures the healing of a pressure ulcer by actually measuring the depth and width, in 2 dimensions, of a wound. A wound heals from the wound bed and closes from the inside to the outside if healthy pink granulation tissue can be seen. This tool contributes to the consistency of measurement of a healing wound.

CONTACTS AND LOCATIONS:
Overall Officials: Cathey Powers, MD, Principal Investigator — Central Arkansas VA/UAMS College of Medicine; Ronni Chernoff, PhD, Principal Investigator — Central Arkansas VA/UAMS College of Medicine
Locations (1):
- Central Arkansas Veterans Healthcare System, Little Rock, Arkansas, United States